CLINICAL TRIAL: NCT00209040
Title: Fear Potentiation and Fear Inhibition in Posttraumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Erica Duncan, MD, Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00000983
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; Acoustic startle
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Subjects with posttraumatic stress disorder
  Interventions: Behavioral: Acoustic Startle Testing
- 2 (Active Comparator): Healthy controls
  Interventions: Behavioral: Acoustic Startle Testing
- 3 (Active Comparator): Combat controls
  Interventions: Behavioral: Acoustic Startle Testing

INTERVENTIONS:
Behavioral: Acoustic Startle Testing — See protocol description for methodological details

SUMMARY:
The current study will investigate the ability of people with and without fear symptoms after trauma to inhibit fear in an experimental situation.

DETAILED DESCRIPTION:
Title of addendum: fear potentiation, conditional discrimination, and fear inhibition in posttraumatic stress disorder.

Principal Investigator: Erica Duncan, M.D.

Co-Investigator: Seth Norrholm, M.D.

Background:

Fear potentiation of the acoustic startle response (ASR) can be demonstrated in both animals and humans (Davis et al., 1993; Grillon et al., 1991). The neural correlates of fear potentiated startle are well studied (Davis et al., 1993) and this paradigm has face validity with cardinal symptoms of posttraumatic stress disorder (PTSD). Central to the clinical problem of PTSD is the inability of these patients to inhibit their fear to stimuli reminiscent of their traumatic experience, even during safe conditions. The elucidation of mechanisms of fear inhibition that may be abnormal in these patients has the potential to advance the development of effective treatments for these patients.

Two conditioning paradigms would permit the study of fear inhibition, but each has potential confounds complicating the interpretation of results. Extinction paradigms have the problem that the same stimulus causes both excitation of the response and later inhibition of response, so that it is difficult to tease apart whether a given experimental manipulation that enhances extinction does so by increasing inhibition or disrupting excitation. Conditioned inhibition (using an A+/AX- paradigm) has the advantage of having two separate stimuli for excitation and inhibition (A is excitatory; X is inhibitory), but has the disadvantage of potential second-order conditioning (i.e., it is possible that A will second-order condition X), which greatly complicates the separation of excitation and inhibition.

The Davis lab has recently developed a discrimination procedure that avoids these problems and allows for the independent evaluation of excitation and inhibition of fear conditioning. The procedure, referred to as a conditional discrimination (abbreviated as AX+/BX-), is based on a paradigm used in earlier learning theory experiments (Rescorla and Wagner, 1972; Bouton and Swartzentruber, 1986). In this experiment, the response to X is conditional upon the presence of either A or B. A becomes excitatory with training as the subject learns that A and X presented together predicts the unconditioned stimulus (US). B becomes inhibitory in that B presented with X predicts safety from the US. The presentation of AB results in a reduced response compared to the response to A alone because B is inhibitory. Accordingly, a novel stimulus, C, paired with A results in a greater response compared to AB. X becomes excitatory to the degree that B is inhibitory. Testing of this paradigm with rats in the Davis lab has produced data in good accord with predicted values (see Figure 1 in Appendix), and does indeed allow for independent evaluation of excitatory and inhibitory processes within the conditioning test session. To date, this paradigm has not been well studied in human subjects. The translation of this paradigm to human subjects would present an important advance in methodology for studying the neurobiology of fear inhibition in clinical populations with anxiety disorders such as PTSD.

Specific Aims:

1. To establish methodology to assess baseline acoustic startle, fear potentiation of acoustic startle in a classical conditioning paradigm, and conditional discrimination (AX+/BX-) in 15 normal control subjects. Fear extinction will be assessed in one to three separate repeated experimental sessions.
2. To compare 15 subjects with PTSD, 15 subjects with a history of combat exposure but no PTSD, and 15 normal controls using this acoustic startle methodology. We hypothesize that PTSD subjects will have normal baseline startle, intact fear potentiation, and impaired inhibition of fear potentiation as measured by the AX+/BX- paradigm. We predict that combat controls will have results intermediate between PTSD subjects and normals.

Methods

Subjects: 75 subjects with PTSD ages 18-80, 75 age and gender matched normal controls, and 75 age and gender matched subjects with combat history but no PTSD will be recruited. Subjects will be screened and excluded for Axis I and II disorders (other than PTSD for the patient group), for significant medical illness, and for auditory or visual impairment.

Assessment: PTSD subjects will be rated for current psychopathology with the Clinician Administered PTSD Scale and the Mississippi Scale for Combat-Related PTSD. In addition, PTSD subjects and combat controls will be rated for severity of combat exposure with the Combat Exposure Scale. In all subjects, childhood trauma will be assessed with the Early Trauma Inventory. Current depression and anxiety symptoms will be assessed using the Hamilton Depression and Hamilton Anxiety scales, respectively. Attention and distractibility will be assessed by means of the Continuous Performance Test, and motor function will be assessed with the Finger Tapping Test. Cognitive function will be assessed with the Benton Visual Retention Test, the California Verbal Learning Test, Wechsler Abbreviated Scale of Intelligence, Wechsler Memory Scale, Selective Reminding Test, and the Trails Test. Results of these tests will be used as covariates in the analysis of conditioning data in order to control for potential group differences in attention or memory. Total time of assessment should be about four to five hours.

Procedure: Acoustic stimuli will be delivered binaurally through headphones (Maico,TDH39P). Acoustic startle stimuli will be 40 ms 116 dB white noise bursts with near instantaneous rise time delivered by a computerized electromyographic (EMG) startle response monitoring system (SR-LAB, San Diego Instruments). The eyeblink component of the acoustic startle response will be measured via EMG of the right orbicularis oculi muscle. EMG activity will be amplified and digitized using the SR-LAB (San Diego Instruments). According to methods established by Davis and Grillon (Grillon et al., 1991; Grillon and Ameli, 1998), aversive stimuli (US) will be 40-250 ms airblasts with an intensity of 100 psi directed to the larynx, emitted by an compressed air tank attached to a polyethylene tubing and controlled by a solenoid switch. A, B, C, and X will be green, purple, orange, or blue lights (counterbalanced color assignment across subjects) or pictures. Subjects will be asked to press a button to indicate that they have learned the discrimination between the different colored lights or pictures. The test session will begin with startle probes to reduce initial startle reactivity and rule out nonstartlers. The training phase of the session will consist of trials in which stimuli A and X are paired with the US (AX+), and trials in which stimuli B and X are not paired with the US (BX-). The test phase will include startle probes alone or during presentation of the cues AB and AC (the order will be counterbalanced across subjects). Between the presentation of AB and AC, there will be reinforced trials of AX. Total time of test session will be approximately 20 minutes.

Statistical Analysis: The basic approach will be a mixed model ANOVA, using Diagnostic Group as a between-subjects factor (for Specific Aim 2), and within-subjects factors of trial type (Cue + Startle vs. Startle Alone), and type of cue (AX, BX, AB, AC).

Future Directions: This work will be coordinated with a series of preclinical studies planned in the Davis lab. The effects of pharmacologic probes on fear conditioning and fear inhibition will be explored in normal controls as a potential method for identifying new pharmacologic treatments for PTSD. Treatment effects on fear conditioning and inhibition will be studied in PTSD subjects. Data from the current project will serve as pilot data for future NIH R01 and VA Merit Review grant submissions.

References:

Bouton ME, Swartzentruber D (1986). Analysis of the associative and occasion-setting properties of contents participating in a Pavlovian discrimination. J Exp Psych Anim Behav Process 12:333-50.

Davis M, Falls WA, Campeau S, Kim M (1993). Fear-potentiated startle: a neural and pharmacological analysis. Behav Brain Res 58:175-98.

Grillon C, Ameli R (1998). Effects of threat and safety signals on startle during anticipation of aversive shocks, sounds, or airblasts. J Psychophysiol 12:329-337.

Grillon C, Ameli R, Woods SW, Merikangas K, Davis M (1991). Fear-potentiated startle in humans: effects of anticipatory anxiety on the acoustic blink reflex. Psychophysiology 28:588-595.

Rescorla RA, Wagner AR (1972). A theory of Pavlovian conditioning: variations in the effectiveness of reinforcement and nonreinforcement. New York: Appleton-Century-Crofts.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Diagnosis of PTSD
* Healthy controls (no history of PTSD)
* Combat controls (no history of PTSD)

Exclusion Criteria:

* No drug or alcohol abuse or dependence

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2001-01; Primary Completion 2012-02-22 (Actual); Study Completion 2012-02-22 (Actual)

PRIMARY OUTCOMES:
Fear potentiation of acoustic startle | Baseline
  Percent change in acoustic startle magnitude during visual cue conditioned to aversive stimuli, compared to trials without aversive stimuli

CONTACTS AND LOCATIONS:
Overall Officials: Erica Duncan, MD, Principal Investigator — Emory University/Atlanta VA Medical Center
Locations (1):
- Atlanta VA Medical Center, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No